CLINICAL TRIAL: NCT06156488
Title: Transcriptome Analysis of Human Bone Regeneration After Using an Anorganic Bovine Bone Graft With or Without a Combination of Polynucleotides and Hyaluronic Acid
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Miguel Padial-Molina, Associate Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0003-N-23
Record Dates: First submitted 2023-11-25; First posted 2023-12-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Sinus Floor Augmentation
MeSH Terms: interventions — Sinus Floor Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anorganic bovine bone (Active Comparator): Maxillary sinus floor augmentation grafted with anorganic bovine bone
  Interventions: Procedure: Maxillary sinus floor augmentation
- Anorganic bovine bone + polynucleotides and hyaluronic acid (Experimental): Maxillary sinus floor augmentation grafted with anorganic bovine bone + polynucleotides and hyaluronic acid
  Interventions: Procedure: Maxillary sinus floor augmentation

INTERVENTIONS:
Procedure: Maxillary sinus floor augmentation — Maxillary sinus floor augmentation through a lateral window grafted with anorganic bovine bone + polynucleotides and hyaluronic acid
  Arms: Anorganic bovine bone + polynucleotides and hyaluronic acid
Procedure: Maxillary sinus floor augmentation — Maxillary sinus floor augmentation through a lateral window grafted with anorganic bovine bone
  Arms: Anorganic bovine bone

SUMMARY:
The goal of this clinical trial is to compare the expression of multiple genes related to bone regeneration in maxillary bone after being grafted with a commonly used biomaterial supplemented or not with a combination of hyaluronic acid and polynucleotides.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients.
* Kennedy class I in the upper jaw.
* Less than 5 mm of residual crestal bone to the maxillary sinus.
* Need for the replacement of teeth with dental implants.

Exclusion Criteria:

* Sinus pathology (sinusitis, mucocele, cysts).
* Smokers.
* Previous long-term (>3 months) use of drugs known to affect bone metabolism, such as bisphosphonates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Transcriptome analysis | 6 months
  Transcriptome analysis of a sample of the regenerated bone will be performed 6 months after grafting immediately before implant placement

SECONDARY OUTCOMES:
Sinus floor height change | 6 months
  CBCT scans will be performed after the sinus floor elevation and 6 months later before implant placement to calculate vertical bone height change

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granada, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Galindo-Moreno P, Abril-Garcia D, Carrillo-Galvez AB, Zurita F, Martin-Morales N, O'Valle F, Padial-Molina M. Maxillary sinus floor augmentation comparing bovine versus porcine bone xenografts mixed with autogenous bone graft. A split-mouth randomized controlled trial. Clin Oral Implants Res. 2022 May;33(5):524-536. doi: 10.1111/clr.13912. Epub 2022 Mar 3. PMID 35224778
- [Background] Galindo-Moreno P, de Buitrago JG, Padial-Molina M, Fernandez-Barbero JE, Ata-Ali J, O Valle F. Histopathological comparison of healing after maxillary sinus augmentation using xenograft mixed with autogenous bone versus allograft mixed with autogenous bone. Clin Oral Implants Res. 2018 Feb;29(2):192-201. doi: 10.1111/clr.13098. Epub 2017 Oct 26. PMID 29071736